CLINICAL TRIAL: NCT07271056
Title: Sublingual Misoprostol Versus No Cervical Priming Before Hysteroscopic Resection of Symptomatic Uterine Niches: Results From a Prospective Randomized Controlled Trial
Brief Title: Sublingual Misoprostol Versus No Cervical Priming Before Hysteroscopic Resection of Symptomatic Uterine Niches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abdel Latif Ahmed Alnezamy, Principal Investigator and Lecturer of Obstetrics and Gynecology, Faculty of Medicine, Benha University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC11-2-2025
Record Dates: First submitted 2025-11-27; First posted 2025-12-08 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Scar Niche; Abnormal Uterine Bleeding; Cesarean Section Complications
Keywords: Misoprostol; Administration, Sublingual; Cervical Priming; Hysteroscopy; Cesarean Section Scar Defect; Randomized Controlled Trial; Postmenstrual Spotting
MeSH Terms: conditions — Metrorrhagia | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Misoprostol group (Active Comparator): Misoprostol group received 200 µg sublingual misoprostol tablet two hours before hysteroscopic resection of uterine niche.
  Interventions: Drug: Misoprostol 200mcg Tab; Procedure: Hysteroscopic resection of uterine niche; Diagnostic Test: Saline-infusion Sonohysterography
- Placebo group (Placebo Comparator): Placebo group received sublingual identical placebo tablet two hours before hysteroscopic resection of uterine niche.
  Interventions: Other: Placebo tab; Procedure: Hysteroscopic resection of uterine niche; Diagnostic Test: Saline-infusion Sonohysterography

INTERVENTIONS:
Drug: Misoprostol 200mcg Tab — Misoprostol group received 200 µg sublingual misoprostol tablet two hours before hysteroscopic resection of uterine niche. A trained nurse, independent of assessment, prepared and administered the medication to the participants.
  Other Names: Misotac®, Sigma Pharmaceutical Industries, Egypt
  Arms: Misoprostol group
Other: Placebo tab — Placebo group received sublingual identical tablet two hours before hysteroscopic resection of uterine niche. A trained nurse, independent of assessment, prepared and administered the tab to the participants.
  Arms: Placebo group
Procedure: Hysteroscopic resection of uterine niche — Procedures were performed around cycle day 10 under spinal or general anesthesia using a 9-mm resectoscope (Karl Storz, Germany) with monopolar energy and 3.5% sorbitol for uterine distension. The Sanders and Murji technique was adapted as follow: (1) anatomical orientation, (2) cephalic rim resection, (3) caudal rim resection, and (4) rollerball ablation of the niche base.
Diagnostic Test: Saline-infusion Sonohysterography — All participants were evaluated by a single blinded sonographer experienced in niche assessment. First, transvaginal ultrasound was performed to exclude pregnancy or pelvic pathology, followed by saline-infusion sonohysterography (2D, sagittal and coronal views). A niche was defined as ≥ 2 mm myometrial indentation at the scar site. Niche depth, length, width, and residual myometrial thickness were recorded.

SUMMARY:
The purpose of the study is to evaluated whether preoperative sublingual misoprostol can enhance the effectiveness and safety of niche resection in patients with symptomatic uterine niche.

DETAILED DESCRIPTION:
After eligibility and consenting, Participants with symptomatic uterine niche were randomized (1:1) to sublingual misoprostol or placebo. Baseline demographic and clinical variables (age, BMI, number of prior cesarean section, number of days of postmenstrual spotting, pelvic pain, dysmenorrhea, dyspareunia, and dysuria) were collected. Symptom severity was assessed using a visual analogue scale (VAS, 1-10). Baseline niche characteristics (residual myometrial thickness, depth, length, and width) were measured by saline infusion sonohysterography. The misoprostol group received 200 µg sublingual misoprostol tablet two hours before surgery; controls received identical placebo tablets. Hysteroscopic resection of uterine niche was performed around cycle day 10 under spinal or general anesthesia using a 9-mm resectoscope with monopolar energy and 3.5% sorbitol for uterine distension. Misoprostol-related adverse events (cramping, fever, GI upset) were recorded preoperatively by a trained nurse. The Sanders and Murji technique was adapted as follow: (1) anatomical orientation, (2) cephalic rim resection, (3) caudal rim resection, and (4) rollerball ablation of the niche base . Intraoperative data (duration, need for dilators, intra- and postoperative complications). At 3 months postoperatively, participants were reassessed for reduction in number of days of postmenstrual spotting, changes in pelvic pain, dysmenorrhea, dyspareunia, and dysuria (VAS scores), participants satisfaction (satisfied/very satisfied vs. dissatisfied/neutral), , and sonohysterographic niche measurements (RMT, depth, length, width).

The participants, hysteroscopist, outcome assessors, and the investigator were blinded for the assignment of the participants to either groups.

ELIGIBILITY:
Inclusion Criteria:

* ≥1 previous cesarean section
* Post cesarean section uterine niche confirmed by saline infusion sonohysterography (niche depth ≥2 mm)
* Residual myometrial thickness ≥2.5 mm as confirmed by saline infusion sonohysterography
* Regular cycles
* Abnormal uterine bleeding for ≥3 consecutive cycles
* Post menstrual spotting or brownish discharge ≥2 days
* Total monthly bleeding duration >7 days

Exclusion Criteria:

* Irregular cycles
* Amenorrhea
* Abnormal cervical cytology
* Acute or chronic cervicitis
* Pelvic inflammatory disease
* Endometrial polyps
* Uterine fibroids
* Contraindications to spinal or general anesthesia
* Refusal to participate

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2025-02-11 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Reduction in number of days of postmenstrual spotting. | At 3 months postoperative.
  The number of days of postmenstrual spotting was recorded at baseline and 3 months post hysteroscopic resection of uterine niche.

SECONDARY OUTCOMES:
Total bleeding days per cycle | At baseline and at 3 months postoperative.
  Total bleeding days per cycle was recorded at baseline and 3 months post hysteroscopic resection of uterine niche.
Pelvic pain score | At baseline and at 3 months postoperative.
  Pain was assessed using a 10-cm Visual Analog Scale (VAS). Participants mark a point on the line that represents their pain,giving that 0 means no pain and 10 means worst pain imaginable. The clinician measures the distance (in centimeters or millimeters) from 0 to the patient's mark and that number is the VAS pain score.
Dysmenorrhea score | At baseline and at 3 months postoperative.
  Pain was assessed using a 10-cm Visual Analog Scale (VAS). Participants mark a point on the line that represents their pain,giving that 0 means no pain and 10 means worst pain imaginable. The clinician measures the distance (in centimeters or millimeters) from 0 to the patient's mark and that number is the VAS pain score.
Dyspareunia score | At baseline and at 3 months postoperative.
  Pain was assessed using a 10-cm Visual Analog Scale (VAS). Participants mark a point on the line that represents their pain,giving that 0 means no pain and 10 means worst pain imaginable. The clinician measures the distance (in centimeters or millimeters) from 0 to the patient's mark and that number is the VAS pain score.
Dysuria score | At baseline and at 3 months postoperative.
  Pain was assessed using a 10-cm Visual Analog Scale (VAS). Participants mark a point on the line that represents their pain,giving that 0 means no pain and 10 means worst pain imaginable. The clinician measures the distance (in centimeters or millimeters) from 0 to the patient's mark and that number is the VAS pain score.
Satisfaction with the outcome | At 3 months postoperative.
  Participant satisfaction with the outcome was assessed using a binary scale (Yes when satisfied/very satisfied , No when dissatisfied/neutral).
Uterine niche measurements | At baseline and at 3 months postoperative.
  First, transvaginal ultrasound was performed to exclude pregnancy or pelvic pathology, followed by saline-infusion sonohysterography (2D, sagittal and coronal views). A niche was defined as ≥ 2 mm myometrial indentation at the scar site. Niche depth, length, width, and residual myometrial thickness were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: AHMED ALNEZAMY, MD, Principal Investigator — Lecturer of Obstetrics and Gynecology, Faculty of Medicine, Benha University
Locations (1):
- Benha Univesity Hospital, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jordans IPM, de Leeuw RA, Stegwee SI, Amso NN, Barri-Soldevila PN, van den Bosch T, Bourne T, Brolmann HAM, Donnez O, Dueholm M, Hehenkamp WJK, Jastrow N, Jurkovic D, Mashiach R, Naji O, Streuli I, Timmerman D, van der Voet LF, Huirne JAF. Sonographic examination of uterine niche in non-pregnant women: a modified Delphi procedure. Ultrasound Obstet Gynecol. 2019 Jan;53(1):107-115. doi: 10.1002/uog.19049. PMID 29536581
- [Background] Zhuo Z, Yu H, Jiang X. A systematic review and meta-analysis of randomized controlled trials on the effectiveness of cervical ripening with misoprostol administration before hysteroscopy. Int J Gynaecol Obstet. 2016 Mar;132(3):272-7. doi: 10.1016/j.ijgo.2015.07.039. Epub 2015 Dec 11. PMID 26797202
- [Background] Tanha FD, Salimi S, Ghajarzadeh M. Sublingual versus vaginal misoprostol for cervical ripening before hysteroscopy: a randomized clinical trial. Arch Gynecol Obstet. 2013 May;287(5):937-40. doi: 10.1007/s00404-012-2652-4. Epub 2012 Dec 4. PMID 23208460
- [Result] Sanders AP, Murji A. Hysteroscopic repair of cesarean scar isthmocele. Fertil Steril. 2018 Aug;110(3):555-556. doi: 10.1016/j.fertnstert.2018.05.032. PMID 30098702
- [Result] Feng YL, Li MX, Liang XQ, Li XM. Hysteroscopic treatment of postcesarean scar defect. J Minim Invasive Gynecol. 2012 Jul-Aug;19(4):498-502. doi: 10.1016/j.jmig.2012.03.010. Epub 2012 May 22. PMID 22621994
- [Result] Nguyen AD, Nguyen HTT, Duong GTT, Phan TTH, Do DT, Tran DA, Nguyen TK, Nguyen TB, Ville Y. Improvement of symptoms after hysteroscopic isthmoplasty in women with abnormal uterine bleeding and expected pregnancy: A prospective study. J Gynecol Obstet Hum Reprod. 2022 Mar;51(3):102326. doi: 10.1016/j.jogoh.2022.102326. Epub 2022 Jan 25. PMID 35091125